CLINICAL TRIAL: NCT04551716
Title: Assessment of Metabolic Associated Fatty Liver Disease (MAFLD) in Chinese Population Using ATI / SWE / SWD: a Prospective Multicenter Study
Brief Title: Noninvasive Assessment of Metabolic Associated Fatty Liver Disease (MAFLD) in Chinese Population
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Principal Investigator, Chinese PLA General Hospital
Other Study IDs: S2020-298-01-01
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Metabolic-dysfunction-associated Fatty Liver Disease (MAFLD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Attenuation imaging (ATI) technology independently developed by Canon medical is a non-invasive examination technology for quantitative detection and analysis of liver steatosis. The technique is simple, rapid and quantitative diagnosis, and is suitable for screening and popularization of early liver steatosis in MAFLD. As noninvasive and effective detection measures of liver inflammation and liver fibrosis, SWD and SWE are more and more widely used in the quantitative diagnosis of liver inflammation and fibrosis. Therefore, ATI combined with SWD / SWE detection can quantitatively diagnose different pathological stages (steatosis, necrotizing inflammation and liver fibrosis) in the development of MAFLD, so as to provide an important basis for treatment.

ELIGIBILITY:
Inclusion Criteria:

1. being a Chinese citizen aged 18 to 85 years;
2. meeting the diagnostic criteria for MAFLD;
3. willing and able to provide informed consent;
4. having a platelet count of at least 50 × 109/L and prothrombin activity of ≥50%.

Exclusion Criteria:

1. The pregnant.
2. Patients who have received or are undergoing systemic chemotherapy.
3. Patients with hepatitis C, alcoholic liver disease (more than 5 years of drinking history, equivalent to alcohol volume ≥ 40g / D in male and ≥ 20g / D in female), drug-induced liver disease or autoimmune hepatitis.
4. Those who re fuse to sign informed consent;
5. There was a significant risk of bleeding (platelet < 50x109 / L, prothrombin activity < 50%).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the results of HBV surface antigen, the patients were divided into two subgroups: (1) HBV surface antigen negative group: pure mafld group; (2) HBV surface antigen positive group: mafld combined with hepatitis B group
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Correlation between ATI / SWD / SWE parameters and the degree of steatosis, inflammation and fibrosis in MAFLD patients | from October 2020 to june 2022

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China